CLINICAL TRIAL: NCT06263777
Title: Nurses Training Program for Early Detection of Children With Developmental Disabilities
Brief Title: Early Detection of Children With Developmental Disabilities in Assiut Governorate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tayseer Saber Younes, Lecturer, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P.T.REC/012/004142
Record Dates: First submitted 2023-11-26; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Developmental Disability; Development Delay; Motor Delay; Down Syndrome; Autism Spectrum Disorder
Keywords: Nurses training; early detection; early intervention; developmental disabilities; children
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities; Psychomotor Disorders; Down Syndrome; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses group (Experimental): Nurse training program on early detection of disability. It included four main elements, which are: a booklet defining different disabilities; a list of the guidelines for early detection; a guide for family guidance for families of children with disabilities; and a monitoring and follow-up form for cases of children with disabilities.
  Interventions: Other: Nurses training program on early detection of disability

INTERVENTIONS:
Other: Nurses training program on early detection of disability — It included four main elements, which are: a booklet defining different disabilities, a list of the guidelines for early detection, a guide for family guidance for families of children with disabilities, a monitoring and follow-up form for 8 cases of children with disabilities). The program consisted of twelve training sessions with a total of 48 hours (4 hours per session) and was based on the techniques of lecture, dialogue, working groups, cooperative learning techniques and participatory learning

SUMMARY:
The study aimed to determine the effectiveness of a designed training program for nurses toward early detection of developmental disabilities among children (0-3 years).

DETAILED DESCRIPTION:
A group of twenty-one licensed nurses with professional experience ranging from 5 to 11 years participated in the study. The participants completed the measurements to evaluate their current knowledge, practice, and perception pre-, post-, and follow-up of the training program in relation to the early detection of disabilities.

ELIGIBILITY:
Inclusion Criteria:

* The study was conducted in selected health units in Assiut, an Upper Egypt Governorate, in selected villages:

  * far from the main government services,
  * without access to public or subsidized transportation to and from the selected villages, and
  * without the presence of any allied health professionals (physical therapists, occupational therapists, speech and language therapists, psychologists), who do not offer any of these medical services.

The selected nurses should be

* employed by the village health department in the public sector,
* locals of the village where the health unit is located,
* and untrained in the early identification or examination of disabled children.

Exclusion Criteria:

* other than inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire of Screening and referral knowledge | 1 month
  percentage of nurses' knowledge about screening and referral of all types of developmental disabilities. minimum score is worst, while maximum is the best
Questionnaire of Disability Perception | 1 month
  The degree of needs of children with developmental delays and the importance of early intervention. minimum score is worst, while maximum is the best
questionnaire about Monitoring Practices | 1 month
  Types of nurses' practices about developmental delay monitoring and assessment.minimum score is worst, while maximum is the best
Follow up | 2 months
  The program's long-term learning effect was measured by the previous outcomes. Minimum score is worst, while maximum is the best

CONTACTS AND LOCATIONS:
Overall Officials: Tayseer S Abdeldayem, PhD, Principal Investigator — Beni-Suef University
Locations (1):
- Tayseer Saber Abdeldayem, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to any other researchers

REFERENCES:
- [Result] Chödrön, G., Pizur-Barnekow, K., Viehweg, S., Puk-Ament, A., & Barger, B. (2019). Childcare providers' attitudes, knowledge, and practice related to developmental monitoring to promote early identification and referral Early Child Development and Care, 1-15. https://doi.org/10.1080/03004430.2019.1626373